CLINICAL TRIAL: NCT06650085
Title: PROtective IleoStomy Versus ProtectivE Colostomy in Anterior Rectal ResectIon - a Multicenter, Open-label, Randomized ConTrolled StudY (PROSPERITY)
Brief Title: Protective Ileostomy Versus Protective Colostomy in Anterior Rectal Resection
Acronym: PROSPERITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Mary and Georg Ehrnrooth's foundation (Unknown); Helsinki University Hospital Research Funds (Unknown)
Responsible Party: Principal Investigator, Ville Sallinen, Adj. Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROSPERITY
Record Dates: First submitted 2024-08-20; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Stoma Colostomy; Stoma Ileostomy
MeSH Terms: interventions — Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loop ileostomy (Experimental)
  Interventions: Procedure: Loop ileostomy
- Loop colostomy (Active Comparator)
  Interventions: Procedure: Loop colostomy

INTERVENTIONS:
Procedure: Loop ileostomy — Patient undergoing anterior rectal resection will receive loop ileostomy
  Arms: Loop ileostomy
Procedure: Loop colostomy — Patient undergoing anterior rectal resection will receive loop colostomy
  Arms: Loop colostomy

SUMMARY:
Loop ileostomy and loop colostomy are both used as protective stomas after anterior resection. There is a lack of evidence on the superiority of loop ileostomy versus loop colostomy. This is a multicenter, open-label, superiority, individually randomized controlled trial including patients undergoing anterior rectal resection with primary anastomosis and a protective stoma. Patients scheduled for anterior rectal resection are randomized 1:1 to loop ileostomy or loop colostomy intraoperatively. Primary outcome is cumulative stoma-related adverse events within 60 days post-primary surgery (scored using Comprehensive Complication Index (CCI)).

ELIGIBILITY:
Inclusion Criteria: Patients undergoing anterior resection (resection of the rectum and colorectal or coloanal anastomosis) due to a rectal tumour and a protective stoma is planned.

The exclusion criteria are: (1) patient already having a stoma (or another stoma made during surgery), (2) technical inability to create ileo- or colostomy (e.g. previous bowel resection, anatomical factors), (3) age <18 years, (4) inadequate ability to co-operate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Stoma-related adverse events | Within 60 days from randomization
  Stoma-related adverse events score by using Comprehensive Complication Index

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days from randomization
  All complications scored using Comprehensive Complication Index
Postoperative complications after stoma closure | Within 30 days from stoma closure
  All complications after stoma closure using Comprehensive Complication Index (including only patients who have undergone stoma closure within 1 year from primary surgery)
Hospital-free days | Within 30 days from randomization
  Days patient is alive and out of any hospital
Quality of life | At 2 months from randomization
  Quality of life measured using EORTC Quality of life questionnaires core 30 with colorectal 29 extension (QLQ-C30+QLQ-CR29)
Kidney function change | Within 1 year from randomization
  Kidney function change defined as difference in eGFR before and 1 year after randomization

OTHER OUTCOMES:
5-year overall survival | Within 5 years from randomization
  Number of patients alive within 5 years from randomization
5-year disease-free survival | Within 5 years from randomization
  Number of patients alive and disease-free within 5 years from randomization (including only patients with M0 at primary operation undergoing radical R0/1 surgery)
Kidney function change at 5 years | Within 5 years from randomization
  Kidney function change defined as difference in eGFR before and 5 years after randomization
Incisional hernia | Within 5 years from randomization
  Number of incision hernias of ostomy site (only patients who have undergone successful stoma closure and alive at 5 years will be included in this analysis)
Stoma closure | Within 5 years from randomization
  Cumulative death-censored successful stoma closure
Quality of life at 5 years | At 5 years from randomization
  Quality of life measured using QLQ-C30 with QLQ-CR29 extension
Quality of life at 5 years | At 5 years from randomization
  Quality of life measured using EQ-5D-5L
Quality of life at 5 years | At 5 years from randomization
  Quality of life measured using low anterior resection syndrome score (LARS scores)
Quality of life at 1 year | At 1 year from randomization
  Quality of life measured using low anterior resection syndrome score (LARS scores)
Quality of life at 6 months | At 6 months from randomization
  Quality of life measured using low anterior resection syndrome score (LARS scores)
Quality of life at 1 year | At 1 year from randomization
  Quality of life measured using EQ-5D-5L
Quality of life at 6 months | At 6 months from randomization
  Quality of life measured using EQ-5D-5L
Quality of life at 2 months | At 2 months from randomization
  Quality of life measured using EQ-5D-5L
Quality of life at 1 year | At 1 year from randomization
  Quality of life measured using QLQ-C30 with QLQ-CR29 extension
Quality of life at 6 months | At 6 months from randomization
  Quality of life measured using QLQ-C30 with QLQ-CR29 extension
Anastomotic leakage | Within 60 days from randomization
  Total number of anastomotic leakages reported also with grading (Rahbari et al., 2010)
Intestinal microbiome | Within 5 years from randomization
  Intestinal microbiome (only patients of the Helsinki University Hospital) composition and functional potential during the stoma in place and stabilization of microbiome after stoma closure.

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koskenvuo L, Paajanen P, Varpe P, Seppala T, Mentula P, Haapamaki C, Carpelan-Holmstrom M, Carpelan A, Lehto K, Satokari R, Lepisto A, Sallinen V. PROtective ileoStomy versus ProtectivE colostomy in anterior Rectal resectIon: study protocol for a multicenter, open-label, randomised conTrolled studY (PROSPERITY). BMJ Open. 2025 May 6;15(5):e096091. doi: 10.1136/bmjopen-2024-096091. PMID 40335149